CLINICAL TRIAL: NCT04447976
Title: A Multi-center Prospective Study to Evaluate Performance of Disposable TIP Duodenoscope Designed to Prevent Future Outbreak Related to Contaminated Duodenoscope.
Brief Title: Prospective Evaluation of Performance of Disposable Elevator Cap Duodenoscope During ERCP in Clinical Practice
Acronym: deCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Wake Forest University Health Sciences (Other); Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-20-0408
Record Dates: First submitted 2020-06-11; First posted 2020-06-25 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: ERCP

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing ERCP by formally trained Endoscopists: No intervention has been used and this is an observational study of evaluation of a TIP duodenoscope performance overall.

SUMMARY:
Purpose: To evaluate overall performance of disposable TIP duodenoscopes and get insight from end-users regarding its performance during various steps of ERCP procedure as well as ease and feasibility of pre-procedure duodenoscope set up and post procedure manual cleaning as well as reprocessing.

Research design: This is a prospective observational multi-center study. Procedure used: During ERCP

Risks and potential benefits: There are no risks associated with this study as it is a retrospective chart review. Potential benefits include the knowledge gained from this study which may be of help to patients in the future.

Importance of knowledge that may reasonably be expected to result: The quality of health care which will be crucial to identify patterns of competence and identify areas of continued improvement. More specifically in the quality metrics sector we will be able to see what is already in place and steps we will undertake that will be beneficial for physicians.

DETAILED DESCRIPTION:
This is a prospective study to evaluate performance of disposable TIP duodenoscopes. Scope is designed to facilitate effective reprocessing of duodenoscope and thus prevent future outbreaks related to contaminated duodenoscope despite standard reprocessing.

This is a multi-center study being performed at the University of Texas Health Science Center, Wake Forest Baptist Health and Institute of Gastroenterology in Ecuador. The study will enroll a total of 100 patients who undergo ERCP. The study is purely observational as it will collect clinical success and information of the TIP duodenoscope.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patients undergoing ERCP.
* Patient has a clinical indication for ERCP.

Exclusion Criteria:

* Any patients less than 18 years old undergoing ERCP as medical necessary procedure.
* Patients who refuse to consent for ERCP procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be outpatients and inpatients undergoing ERCP at the Memorial Hermann Hospital Texas Medical Center. All patients will be seen by any one of the investigators either in the outpatient clinic or during inpatient consultation on hospitalized patients.
  The physicians and Nurse technicians will be evaluating the performance of the TIP duodenoscope on these patients undergoing ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Disposable TIP duodenoscope survey evaluation performance | During procedure
  To evaluate overall performance of disposable TIP duodenoscope through a survey regarding its performance during various steps of ERCP procedure.
To get insight from end-users such as physicians, fellows in training and nurse technicians regarding the disposable TIP duodenoscope performance during various steps of ERCP procedure through a questionnaire provided. | during procedure
  To evaluate overall performance of disposable TIP duodenoscopes through a survey and get insight from end-users such as physicians, fellows in training and nurse technicians regarding its performance during various steps of ERCP procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Thosani, MD, MHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States